CLINICAL TRIAL: NCT05443295
Title: Improvement of Fatigue in Unstable Shoulder Through a Therapeutic Exercise Program in Physiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: Instituto de Investigacion Biomedica de Malaga (Other); Queensland University of Technology (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Physiotherapist. PhD. Professor Department of Physiotherapy, Faculty of Health Sciences, University of Malaga, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MoveUS
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-07

CONDITIONS: Instability, Joint; Shoulder Dislocation; Fatigue; Therapeutic Alliance
Keywords: instability; shoulder; fatigue; exercise
MeSH Terms: conditions — Joint Instability; Shoulder Dislocation; Fatigue; Motor Activity

STUDY DESIGN:
Intervention Model Description: A single-blind randomized controlled trial.
Who Masked: Investigator
Masking Description: An external physiotherapist will be used to supervise the intervention carried out, so that the evaluator does not know at any time which group each subject belongs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will carry out the MoveUS Program.
  Interventions: Other: MoveUS Program
- Control Group (Active Comparator): The control group will be subjected to the conventional guidelines in the approach to shoulder instability.
  Interventions: Other: Control intervention

INTERVENTIONS:
Other: MoveUS Program — The MoveUS Program have 5 stages: 1 (approach stage), based on analytical movements, isometric peak contractions and learning/motor control; 2 (structural stage), based on muscular strength or resistance training through a cumulative work of short efforts, following with the analytical work of pushing or lifting/pulling; and ending in a closed kinetic chain; 3 (neural stage), that has two stage: 3A, based on a structural work that serves as a continuation of stage 2 and the work is focused on the training of increase cross-sectional muscular area; and 3B, based on a neural work focursed in an intra neuromuscular system highlighted motoneuron unit workout. Finally, stage 4 (functional stage), based on a functional readaptation to sports activity and/or work activity; or, failing that, to the activity of daily life with the highest demand.
  Arms: Intervention Group
Other: Control intervention — The control intervention is based on following the conventional treatment guidelines for glenohumeral instability, where immobilization, taking non-steroidal anti-inflammatory drugs, cryotherapy, passive kinesitherapy and self-assisted, pendular exercises stand out and education.
  Arms: Control Group

SUMMARY:
Background: Glenohumeral instability is a highly prevalent pathology; however, there is great controversy in its definition. Traditionally, structural problems such as labral injury or bone loss in the glenoid cavity were considered the main causes; but recently, it has been seen that motor control plays a very relevant role. This means that currently, there is a disparity of action protocols and the treatment of this pathology is a great challenge.

Aim: The primary aim of this study is to evaluate the effectiveness of a supervised multicomponent therapeutic exercise program in reducing multivariable fatigue in patients with instability of the glenohumeral joint.

Methods: A single-blind randomized controlled trial will be carried out, in which 108 adult patients who have suffered at least one episode of glenohumeral instability in the last year will be recruited, who will be randomized to the intervention group, which will carry out a multicomponent therapeutic exercise program supervised by physiotherapists (MoveUS Program); or to the control group, which will receive the usual care. All subjects will be evaluated at baseline, mid-treatment and at the end. In these evaluations, range of movement, maximum peak of isometric force, kinematic, physiological and psychometric fatigue, return to activity, motor control and number of recurrences will be assessed; as well as the quality of life measured through the Western Ontario Shoulder Instability Index, which will be the main outcome variable. A multivariate analysis will be performed through a statistical program.

Discussion: This study aims to determine if therapeutic exercise supervised by physiotherapists is capable of reducing multivariable fatigue, reducing the number of recurrences and improving quality of life; to be able to implement it in the future in public and private centers.

DETAILED DESCRIPTION:
The glenohumeral joint presents a high incidence of dislocation (15.3 - 56.3 per 100,000 people per year), which is often accompanied by injury to the glenoid labrum, which increases the number of patients with chronic glenohumeral instability. However, there is great controversy when it comes to giving a clear and agreed definition among experts, since the term "recurrent glenohumeral instability" has been used in the scientific literature to encompass a multitude of terms such as dislocation, subluxation, apprehension and instability.

The two common points found in most definitions are discomfort and excessive translation of the humeral head in the glenoid fossa.

Traditionally, biomechanics have attributed glenohumeral instability to structural defects, pointing to bone loss in the glenoid cavity and Hill-Sachs lesion as its main causes. Nonetheless, it has been shown that abnormal muscle activation patterns of the periarticular muscles of the shoulder may be the cause of said instability without the need for there is structural damage.

Taking this last clarification into account, in 2020 a consensus was reached among various experts in the field of shoulder surgery to establish a standard in the classification of functional shoulder instability (FSI), dividing it into two large groups defined as positional FSI, when the shoulder subluxation or dislocation occurs during arm movement and is reduced when returning to neutral position; and non-positional FSI, when this glenohumeral dislocation occurs with the shoulder in a neutral position.

Additionally, a subdivision is made based on the patient's ability to control the occurrence of the event: the controllable ones, when the subject is capable of producing and reducing the dislocation voluntarily, almost without symptoms; and uncontrollable when the episode of instability occurs involuntarily, causing more severe pain and functional impotence.

In a more detailed analysis of individuals suffering from functional shoulder instability, electromyography found increased activity in the muscles that stabilize the humeral head and decreased activity in those responsible for mobility. Likewise, a decrease in superointernal scapular rotation was found during arm elevation, generating a descent of the humeral head, which is increased if it is accompanied by ligament hyperlaxity.

The lack of glenohumeral stability can generate a wide variety of signs and symptoms such as pain, limited range of motion, loss of strength, kinesiophobia and a continuous sensation of instability. Added to all this is fatigue, whose early detection can play a very relevant role in the prevention of shoulder injuries, but its evaluation is a great challenge since the term fatigue encompasses several variables.

The kinematic variable refers to both the lack of stability to raise the upper limb and the loss of movement speed. The monitoring of the speed during the execution of the entrusted task can be useful to estimate the number of repetitions that the patient can perform before muscle failure appears.

The physiological variable refers to the inability to generate adenosine triphosphate (ATP) to maintain a movement over time. This insufficiency of metabolic substrate is usually the cause of the so-called neuromuscular fatigue, which has two main axes, central fatigue and peripheral fatigue.

The psychometric variable can manifest itself at the behavioral level, with a decrease in precision in the work carried out; and on a psychological level, with a feeling of exhaustion, weakness and demotivation. This generates an overestimation of the perception of effort and, ultimately, a reduction in physical performance.

In addition to the differentiation of these three variables, when addressing the problem of fatigue, it must be taken into account that there are significant differences related to age and sex.

Taking these findings as a reference, and emphasizing the fact that fatigue is capable of altering the role of the static and dynamic stabilizers of the humeral head, there are already several studies that suggest the need to analyze it in greater depth and establish agreed prevention and rehabilitation protocols in relation to glenohumeral instability.

Exercise plays a fundamental role in this pathology, both in the conservative approach, which is usually the first choice, and in rehabilitation after the surgical approach; since it has been proven that a therapeutic exercise program optimizes the function of dynamic stabilizers that are essential in the maintenance of glenohumeral stability.

In the conservative approach, the Watson program focuses on gaining motor control and stability in the glenohumeral and scapulothoracic joints; and presents six stages that progress over 12 weeks with the strengthening of the axioscapular muscles, the rotator cuff and the deltoid, until the patient is included in their activities of daily living and sports.

This intervention has shown significant improvements compared to other programs such as the Rockwood in the Western Ontario Shoulder Instability Index, in the reduction of pain, in flexor strength and in scapular coordination.

Within this non-surgical approach, the SINEX program is based on 12 weeks of neuromuscular exercises supervised by a physiotherapist with a progression through 7 levels in which strength, coordination, balance and proprioception, as well as the integration of these patterns in functional activities. This intervention reported significant improvements compared to other interventions such as the HOMEX program, especially in apprehension and in the ability to perform sports activities.

Additionally, the influence of the 12-week WIP1 conservative exercise program, through teleconsultation, on atraumatic shoulder instability was analyzed. This program has 6 stages that go through gaining scapular motor control, toning the periarticular muscles, controlling the different planes of movement and integrating movement patterns into specific individualized tasks; reporting significant improvements in stability, shoulder function, strength and scores on specific questionnaires.

When the conservative approach is not successful, there is some trauma in the clinical history or there are concomitant injuries such as Hill-Sachs or Bankart, arthroscopic surgical techniques are used, consisting of the reduction of the joint capsule, since it has been shown that report better long-term results and a lower incidence of recurrence.

After surgery, early supervised mobilization of the involved joint is necessary to optimize the results of the intervention, minimize pain, maximize range of motion and return to sports activity.

The fact of betting on accelerated rehabilitation, in which the patient is subjected to strength and proprioception training with a high demand for skills, to increase precision in stability and joint position, makes it necessary for the exercise program treatment is supervised by a qualified professional in the area.

According to the American Association of Shoulder and Elbow Therapists, rehabilitation after capsulolabral shoulder repair arthroscopy consists of three phases. The first phase focuses on the maximum protection of the surgical sutures. The second phase focuses on achieving functional joint range, submaximal strength, and dynamic stabilization; and the third phase is based on improving neuromuscular function, increasing strength, maximizing joint range and returning the patient to their daily activities and sports practice.

The current challenge in this field is to design an individualized therapeutic exercise program that takes into account the differences in the initial factors between the different individuals, the union between the reduction of symptoms and the return to work and/or sports activity, individual potential, and the conjunction between the protection of tissues and the maximization of capacities; in order to optimize the results of the recovery.

For these reasons, the main objective of this study is to evaluate the effectiveness of a supervised multicomponent therapeutic exercise program in reducing multivariable fatigue in patients with instability of the glenohumeral joint.

ELIGIBILITY:
Inclusion Criteria:

* Having suffered at least one episode of glenohumeral instability in the last year.
* Age between 18 and 64 years.
* Have signed the informed consent.
* Score equal to or less than 6 on the Instability Severity Index Score.

Exclusion Criteria:

* Ethical or cultural barriers.
* Lack of command of Spanish language.
* Underlying diseases or concomitant treatments that may affect exercise capacity.
* Participation in other clinical trials.
* Score equal to or greater than 1800 on the Western Ontario Shoulder Instability Index.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-03-09 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Quality of life (WOSI) | 12 weeks
  Quality of life is the set of factors that contribute to a person's well-being. It will be assessed through the Western Ontario Shoulder Instability Index

SECONDARY OUTCOMES:
Range of movement (ROM) | 12 weeks
  ROM corresponds to the difference in active and passive joint amplitude, measured with the G-pro smartphone application.
Scapulo-humeral rhythm (ECH) | 12 weeks
  The scapulo-humeral rhythm refers to the motor control capacity of the axioscapular and periarticular muscles of the shoulder to perform the movements of the shoulder joint complex, and will be measured through bipolar surface electromyography
Kinematic fatigue (Fc) | 12 weeks
  Kinematic fatigue refers to the loss during the execution of a movement, and will be assessed with inertial sensors and 3D motion capture system.
Physiological fatigue (Ff) | 12 weeks
  Physiological fatigue refers to the inability to produce adenosine triphosphate to support aerobic and anaerobic efforts; and will be evaluated through high density surface electromyography.
Psychometric fatigue (Fp) | 12 weeks
  Psychometric fatigue translates into a decrease in performance, caused by a feeling of exhaustion, weakness and demotivation. It will be assessed with the Quick Piper Fatigue scale-revised.
Maximum peak of isometric force (FIM) | 12 weeks
  Peak isometric force refers to the maximum voluntary force applied when resistance is insurmountable. It will be quantified with an electromechanical dynamometer.
Return to play (RTP) | 12 weeks
  Return to play is characterized by a person's ability to return to their work and sports routine. It will be evaluated with the "Cuestionario sobre la autopercepción del deportista para la reincorporación al entrenamiento normalizado tras una lesión".
Number of recurrences (Nº REC) | 12 weeks
  The number of recurrences is defined as the number of times the patient suffers from the phenomenon of interest again. It will be recorded through an individualized diary.
Glenohumeral stability (STAB) | 12 weeks
  Functional stability of the glenohumeral joint can be defined as the maintenance of the alignment of the center of the humeral head within the glenoid fossa during movement, achieved through the precise probing of static (passive) and dynamic (active) mechanisms; and will be measured with MoveUS Test.
Muscular fatigue (Mf) | 12 weeks
  Muscle fatigue is, in short, muscle fatigue and occurs when there is extreme exhaustion of muscle fibers due to intense physical activity; and will be measured with Modified T-Fast Test.

CONTACTS AND LOCATIONS:
Overall Officials: Cuesta Vargas A Antonio Ignacio, PhD, Principal Investigator — University of Malaga
Locations (2):
- Spain (2):
  - Antonio Cuesta Vargas, Málaga, Málaga
  - Hospital Comarcal de la Axarquía, Málaga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez-Perez L, Cuesta-Vargas AI. Shoulder Muscle Activity Through Surface Electromyography and Estimation of Physiological Fatigue Using the T-Fast Test in Patients With Glenohumeral Instability: A Cross-Sectional Study. Physiother Res Int. 2025 Jul;30(3):e70085. doi: 10.1002/pri.70085. PMID 40543070
- [Derived] Ramirez-Perez L, Cuesta-Vargas AI. Effect of a multicomponent exercise program focused on multivariable fatigue improvement versus standard care for glenohumeral instability: MoveUS study protocol. BMC Musculoskelet Disord. 2024 Dec 18;25(1):1013. doi: 10.1186/s12891-024-08193-4. PMID 39695629